CLINICAL TRIAL: NCT01826747
Title: Impact of Luteal Phase Support With Vaginal Progesterone on the Clinical Pregnancy Rate in Intrauterine Insemination Cycles Stimulated With Gonadotrophins: a Prospective Randomized Multicentre Study.
Brief Title: Intrauterine Insemination and Luteal Fase Support
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S52775
Record Dates: First submitted 2013-02-25; First posted 2013-04-08 (Estimated); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Infertility
Keywords: intrauterine insemination; luteal phase; gonadotrophins
MeSH Terms: conditions — Infertility | interventions — Crinone; Progesterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental (Experimental): Luteal Phase support
  Interventions: Drug: crinone (progesterone 8%, vaginal application)
- control (No Intervention): No luteal Phase support

INTERVENTIONS:
Drug: crinone (progesterone 8%, vaginal application)
  Arms: experimental

SUMMARY:
The objective is to test the hypothesis that luteal phase support with vaginal progesterone leads to a higher clinical pregnancy rate (primary outcome) and live birth rate (secondary outcome) when compared to no luteal phase support in a program of intrauterine insemination (IUI) after controlled ovarian stimulation with gonadotrophins. Additionally, the length of the luteal phase will be recorded (secondary outcome) in order to detect luteal phase defects/insufficiencies in the absence of luteal phase suppletion as well as luteal phase prolongation in case of luteal phase support which may be a burden for the patients waiting for the outcome of the treatment.

ELIGIBILITY:
Inclusion Criteria:

Patients with an indication for IUI:

* unexplained infertility
* mild male factor infertility
* minimal-mild endometriosis

Women:

* first IUI cycle ever
* normal ovulatory cycles (26-32d)
* age<43,BMI≤30
* presence of at least one patent tube on hysterosalpingography and/or laparoscopy
* normal uterine cavity (ultrasound, hysterosalpingography, or laparoscopy)

Men: Total motile count ≥ 5 Million/ml after capacitation

Exclusion Criteria:

* Patients with contra-indication for pregnancy , infertility or progesterone use.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 393 (Actual)
Dates: Start 2011-04 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
clinical pregnancy rate per IUI cycle | by ultrasound at ± 5 to 6 weeks after IUI

SECONDARY OUTCOMES:
live birth rate per IUI cycle | 40 weeks after IUI

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium

REFERENCES:
- [Derived] Peeraer K, D'Hooghe T, Laurent P, Pelckmans S, Delvigne A, Laenen A, Welkenhuysen M, Wyns C, De Neubourg D. Impact of luteal phase support with vaginal progesterone on the clinical pregnancy rate in intrauterine insemination cycles stimulated with gonadotropins: a randomized multicenter study. Fertil Steril. 2016 Nov;106(6):1490-1495. doi: 10.1016/j.fertnstert.2016.07.1096. Epub 2016 Aug 23. PMID 27565253